CLINICAL TRIAL: NCT06036173
Title: Effects of Lymphedema After Breast Cancer Treatment on Body Awareness and Upper Extremity Functionality
Brief Title: Body Awareness and Functionality in Lymphedema
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assist. Prof., Selcuk University
Other Study IDs: 2023/09.06
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Lymphedema of Upper Limb

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- developed lymphedema after breast cancer surgery
  Interventions: Other: diagnosis of lymphedema; Other: breast cancer surgery
- did not develop lymphedema after breast cancer surgery
  Interventions: Other: breast cancer surgery
- without a history of any cancer surgery

INTERVENTIONS:
Other: diagnosis of lymphedema — being diagnosed with secondary lymphedema in the upper extremity according to the International Lymphedema Association
  Groups: developed lymphedema after breast cancer surgery
Other: breast cancer surgery — be diagnosed and undergo surgery
  Groups: developed lymphedema after breast cancer surgery; did not develop lymphedema after breast cancer surgery

SUMMARY:
To determine whether body awareness and upper extremity functionality are affected in patients with or without lymphedema development after breast cancer surgery in comparison with individuals without a history of cancer.

ELIGIBILITY:
Inclusion Criteria:

first group:

* being female,
* being aged 18-65 years,
* having undergone unilateral breast cancer surgery,
* being diagnosed with secondary lymphedema in the upper extremity according to the International Lymphedema Association
* not having any orthopedic disease that would prevent walking, and volunteering to participate in the study.

second group:The inclusion criteria for the breast cancer surgery group

* without lymphedema were being female,
* being aged 18-65 years,
* having undergone unilateral breast cancer surgery, and volunteering to participate in the study.

Lastly, the inclusion criteria for the control group were:

* being female,
* being aged 18-65 years,
* having no history of cancer surgery, and volunteering to participate in the study.

Exclusion Criteria: for all groups

* not being willing to participate in the study;
* the presence of metastases, neurological, or orthopedic disorders;
* postural deformities, such as scoliosis and kyphosis;
* mental and cognitive disorders; or communication/cooperation problems

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: being a woman and having had breast cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnaire | 17 minutes
  This instrument consists of a total of 18 items evaluated based on a scale of 1 (not at all true of me) to 7 (very true of me). The total score is obtained by adding the scores of each item. A higher total score indicates better body awareness. Max/ min score:126/18
Quick-Disabilities of the Arm, Shoulder, and Hand questionnaire | 11 minutes
  Each of the 11 items in this instrument is scored from 1 to 5. The responses given to all items are summed up, and the total score is obtained with a special formula. A high total score indicates a high level of functional limitation. Max/ min score: 100/0

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)